CLINICAL TRIAL: NCT03506620
Title: The Role of Nerve Blocks in Hip Arthroscopy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unforeseen cost restrictions of the drug halted the execution of this study altogether.
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Thomas Lynch, Assistant Professor of Orthopedic Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAR7247
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Femoroacetabular Impingement
Keywords: femoroacetabular impingement; hip arthroscopy; QL nerve block
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Ropivacaine; Saline Solution; Injections

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled, double-blind trial. Patients undergoing hip arthroscopy who agree to participate will be randomly selected to receive an ultrasound-guided QL block with either local anesthetic (QL block group) or normal saline (control group) preoperatively.
Who Masked: Participant, Care Provider
Masking Description: The anesthesiologist, surgeon, and patient will all be blinded to the intervention. After patients consent to join the study, a member of the study team who is not involved in patient care will randomly allocate patients to 1 of 2 groups, the intervention or the controls. A statistician not involved with the study will creat a randomization table and coordinate with the Research Pharmacy to keep the study team blinded. Naropin (Ropivacaine) will be dispensed by the research pharmacy. The nurse will prepare the study injection accordingly for the blind anesthesiologist to administer. The QL block will be administered by a trained musculoskeletal regional anesthesia specialist before the standard induction of general anesthesia. The injection will occur under sedation to minimize discomfort for the patient. The QL block group's injection will consist of 20 cc of 0.25% Ropivacaine, whereas the control group will receive 20 cc of saline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Subjects will be randomized to receive a single-injection QL block with normal saline (Saline Solution for Injection).
  Interventions: Drug: Saline Solution for Injection
- QL Block (Experimental): Subjects will be randomized to receive a single-injection QL block with either local anesthetic (0.25% Ropivacaine injection).
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — Naropin (Ropivacaine HCl) 0.25%; Dose: 20 cc
  Other Names: Naropin
  Arms: QL Block
Drug: Saline Solution for Injection — 20 cc of saline will be injected in the form of a QL block as a placebo.
  Other Names: Normal Saline
  Arms: Control

SUMMARY:
The goal of this study is to determine whether QL blocks reduce opioid consumption following arthroscopic hip surgery by decreasing postoperative pain. Considering the current opioid epidemic, the responsibility of physicians to help prevent addiction, and the increasing prevalence of arthroscopic hip surgeries, this study holds a tremendous potential benefit for future patients.

DETAILED DESCRIPTION:
The popularity of arthroscopic hip surgery has increased greatly over the last 10 years, particularly for correcting Femoroacetabular Impingement (FAI). FAI is a structural abnormality of the proximal femur, the acetabulum, or both. It is a leading cause of labral tears in the hip joint and can cause cartilage damage, which may increase subsequent risk of developing osteoarthritis. Though far less invasive than open hip surgery such as for a total hip replacement, hip arthroscopy can cause significant postoperative pain for the patient. Given how relatively new the procedure still is, methods of pain control are highly variable. Peripheral nerve blocks, mainly femoral nerve and lumbar plexus blocks, have been used by some surgeons to control postoperative pain. However, in addition to their sensory effects, these blocks cause motor impairment that has been associated with a significantly higher risk of falling.

In managing pain after any operation, opioid consumption is, of course, a significant concern. Ideally, hip arthroscopy patients could receive a peripheral nerve block that decreases pain and the need for opioids, but without the muscular weakness and increased fall risk observed with femoral nerve and lumbar plexus blocks. This may be achievable with the newer Quadratus Lumborum (QL) block.

The ultrasound-guided QL block is currently most commonly used for abdominal surgery.

However, several case studies of a single-injection QL block in hip replacement surgeries have been successful in minimizing pain and opioid use while sparing motor function and avoiding the muscle weakness that can lead to falls. In the approach utilized in these cases, local anesthetic was injected at the anterolateral border of the QL muscle to achieve analgesia ranging from the T6-T10 through L3 dermatomes. One group has anecdotally reported great success in using these QL blocks for alleviating postoperative pain with hip arthroscopy, but no studies to date have evaluated the effectiveness of QL blocks for arthroscopic hip surgery.

This study is a randomized, controlled, double-blind trial. Patients undergoing hip arthroscopy who agree to participate will be randomly selected to receive an ultrasound-guided QL block with either local anesthetic (QL block group) or normal saline (control group) preoperatively.

After surgery and during the first postoperative week, patients will record their numerical pain score, the location of their pain, and their opioid consumption using our attached study instrument. On this form, they will record their pain score at 0.5, 1, 1.5, 2, 4, 6, 12, 24, and 48 hours and 7 days after surgery. The form specifies that if patients are unable to record their pain score at any of these time points, particularly because they are sleeping/recovering, they can simply skip that time point. For pain location, patients are instructed to draw X's on a standard cartoon at the site of their pain. For opioid consumption, patients simply record when and how many pills they take. This form will be collected from patients at their 10-14 day postoperative visit. Data will also be collected from the medical chart on time to discharge and any complications in the perioperative period. Questionnaires will be used to assess pain, physical and social health, such as Patient-Reported Outcomes Measurement Information System (PROMIS).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to receive unilateral arthroscopy hip surgery at Columbia University Medical Center with Dr. Lynch.

Exclusion Criteria:

* Patients scheduled to receive bilaterally or staged hip arthroscopy.
* Patients unwilling to participate in the research.
* History of chronic opioid use.
* Contraindication or allergy to study medications, such as QL block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Pain Score | 0.5 hour
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 1 hour
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 1.5 hours
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 2 hours
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 4 hours
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 6 hours
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 12 hours
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 24 hours
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 48 hours
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Pain Score | 7 days
  Patients will record their numerical pain score on a scale of 0 to 10 (0 = no pain, 10 = worst pain imaginable)
Oral Morphine Equivalents | 24 hours after surgery
  Opioid consumption following surgery as self reported by patients, measured in mg
Oral Morphine Equivalents | 48 hours after surgery
  Opioid consumption following surgery as self reported by patients, measured in mg
Oral Morphine Equivalents | 7 days after surgery
  Opioid consumption following surgery as self reported by patients, measured in mg
Patient Satisfaction Score | 24 hours after surgery
  Patients will record their satisfaction following surgery on a scale of 0-10 (0 being not satisfied, 10 being fully satisfied)
Patient Satisfaction Score | 48 hours after surgery
  Patients will record their satisfaction following surgery on a scale of 0-10 (0 being not satisfied, 10 being fully satisfied)
Patient Satisfaction Score | 7 days after surgery
  Patients will record their satisfaction following surgery on a scale of 0-10 (0 being not satisfied, 10 being fully satisfied)
Percentage of Patients Reporting Nausea and/or Vomiting | 24 hours after surgery
  Patients will self report any instances of nausea and/or vomiting
Percentage of Patients Reporting Nausea and/or Vomiting | 48 hours after surgery
  Patients will self report any instances of nausea and/or vomiting
Percentage of Patients Reporting Nausea and/or Vomiting | 7 days after surgery
  Patients will self report any instances of nausea and/or vomiting

SECONDARY OUTCOMES:
HOS-ADL Questionnaire Score | Baseline preoperative
  Hip Outcome Survey (HOS) is a self-administered questionnaire with a scoring system composed of 2 sub-scales - a rating tool to assess a patient's level of ability. Activities of Daily Living (ADL) sub-scale made of 19 items. Scales are scored from 0 to 4, with 0 being 'unable to do' and 4, 'no difficulty'. The average of the total scores of the patients in each arm will be provided.
HOS-ADL Questionnaire Score | 2 weeks after surgery
  Hip Outcome Survey (HOS) is a self-administered questionnaire with a scoring system composed of 2 sub-scales - a rating tool to assess a patient's level of ability. Activities of Daily Living (ADL) sub-scale made of 19 items. Scales are scored from 0 to 4, with 0 being 'unable to do' and 4, 'no difficulty'. The average of the total scores of the patients in each arm will be provided.
mHHS Questionnaire Score | Baseline preoperative
  Modified Harris Hip Score (mHHS) is made up of 8 questions - a rating tool to assess how you are doing before and after surgery. The score is reported as 90-100 for excellent results, 80-89 being good, 70-79 fair, 60-69 poor, and below 60 a failed result.The average of the total scores of the patients in each arm will be provided.
mHHS Questionnaire Score | 2 weeks after surgery
  Modified Harris Hip Score (mHHS) is made up of 8 questions - a rating tool to assess how you are doing before and after surgery. The score is reported as 90-100 for excellent results, 80-89 being good, 70-79 fair, 60-69 poor, and below 60 a failed result.The average of the total scores of the patients in each arm will be provided.
HOOS - Symptoms and Stiffness Questionnaire Score | Baseline preoperatively
  A 40 item questionnaire (hip disability and osteoarthritis outcome score, HOOS) to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included. The average of the total scores of the patients in each arm will be provided.
HOOS - Symptoms and Stiffness Questionnaire Score | 2 weeks after surgery
  A 40 item questionnaire (hip disability and osteoarthritis outcome score, HOOS) to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included. The average of the total scores of the patients in each arm will be provided.
HOOS - ADL Questionnaire Score | Baseline preoperatively
  A 40 item questionnaire (hip disability and osteoarthritis outcome score, HOOS) to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included.This subscale: Activities of Daily Living. The average of the total scores of the patients in each arm will be provided.
HOOS - ADL Questionnaire Score | 2 weeks after surgery
  A 40 item questionnaire (hip disability and osteoarthritis outcome score, HOOS) to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included.This subscale: Activities of Daily Living. The average of the total scores of the patients in each arm will be provided.
HOOS - Sports Questionnaire Score | Baseline preoperatively
  HOOS will be used to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included. This subscale: Sport and Recreation Function (SP) (four items). The average of the total scores of the patients in each arm will be provided.
HOOS - Sports Questionnaire Score | 2 weeks after surgery
  HOOS will be used to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included. This subscale: Sport and Recreation Function (SP) (four items). The average of the total scores of the patients in each arm will be provided.
HOOS - Quality of Life Questionnaire Score | Baseline preoperatively
  HOOS will be used to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included. This subscale: Hip Related Quality of Life (Q) (four items). The average of the total scores of the patients in each arm will be provided.
HOOS - Quality of Life Questionnaire Score | 2 weeks after surgery
  HOOS will be used to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included. This subscale: Hip Related Quality of Life (Q) (four items). The average of the total scores of the patients in each arm will be provided.
UCLA Activity Score Questionnaire Score | Baseline preoperatively
  University of California, Los Angeles (UCLA) activity scale is a simple scale ranging from 1 to 10. The patient indicates her or his most appropriate activity level, with 1 defined as "no physical activity, dependent on others" and 10 defined as "regular participation in impact sports." The average of the total scores of the patients in each arm will be provided.
UCLA Activity Score Questionnaire Score | 2 weeks after surgery
  University of California, Los Angeles (UCLA) activity scale is a simple scale ranging from 1 to 10. The patient indicates her or his most appropriate activity level, with 1 defined as "no physical activity, dependent on others" and 10 defined as "regular participation in impact sports." The average of the total scores of the patients in each arm will be provided.
VR-12 Mental Health Questionnaire Score | Baseline preoperatively
  Veterans Rand 12 Item Health Survey (VR-12) is a brief, generic, multi-use, self-administered health survey comprised of 12 items. The instrument is primarily used to measure health-related quality of life, to estimate disease burden and to evaluate disease-specific benchmarks with other populations. The 12 items are summarized into two scores, one for mental health and one for physical health. The average of the total scores of the patients in each arm will be provided.
VR-12 Mental Health Questionnaire Score | 2 weeks after surgery
  Veterans Rand 12 Item Health Survey (VR-12) is a brief, generic, multi-use, self-administered health survey comprised of 12 items. The instrument is primarily used to measure health-related quality of life, to estimate disease burden and to evaluate disease-specific benchmarks with other populations. The 12 items are summarized into two scores, one for mental health and one for physical health. The average of the total scores of the patients in each arm will be provided.
VR-12 Physical Health Questionnaire Score | Baseline preoperatively
  VR-12 will be used to measure health-related quality of life, to estimate disease burden and to evaluate disease-specific benchmarks with other populations. The 12 items are summarized into two scores, one for mental health and one for physical health.The average of the total scores of the patients in each arm will be provided.
VR-12 Physical Health Questionnaire Score | 2 weeks after surgery
  VR-12 will be used to measure health-related quality of life, to estimate disease burden and to evaluate disease-specific benchmarks with other populations. The 12 items are summarized into two scores, one for mental health and one for physical health.The average of the total scores of the patients in each arm will be provided.
HOOS - Short Form Total Score Questionnaire Score | Baseline preoperatively
  HOOS will be used to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included. The average of the total scores of the patients in each arm will be provided.
HOOS - Short Form Total Score Questionnaire Score | 2 weeks after surgery
  HOOS will be used to assess patient-relevant outcomes in five separate subscales. To answer each question, five Likert-boxes were used (no, mild, moderate, severe, extreme). All items were scored from zero to four, and each of the five subscales was calculated as the sum of the items included. The average of the total scores of the patients in each arm will be provided.
iHOT-12 Questionnaire Score | Baseline preoperatively
  A Short Version of the International Hip Outcome Tool (iHOT-12) self administered outcome measure based on a Visual Analogue Scale response format designed for young and active population with hip pathology. The average of the total scores of the patients in each arm will be provided.
iHOT-12 Questionnaire Score | 2 weeks after surgery
  A Short Version of the International Hip Outcome Tool (iHOT-12) self administered outcome measure based on a Visual Analogue Scale response format designed for young and active population with hip pathology. The average of the total scores of the patients in each arm will be provided.
PROMIS v1.1 Pain Interference Questionnaire Score | Baseline preoperatively
  PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health. The Pain Interference Questionnaire is comprised of 56 items, total score will be calculated. PROMIS is a computer adaptive test with branching logic. To answer each question, five Likert-boxes were used. The average of the total scores of the patients in each arm will be provided.
PROMIS v1.1 Pain Interference Questionnaire Score | 2 weeks after surgery
  PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health. The Pain Interference Questionnaire is comprised of 56 items, total score will be calculated. PROMIS is a computer adaptive test with branching logic. To answer each question, five Likert-boxes were used. The average of the total scores of the patients in each arm will be provided.
PROMIS v1.0 Pain Intensity 3a Questionnaire Score | Baseline preoperatively
  PROMIS is a computer adaptive test with branching logic. The Pain Intensity Questionnaire is comprised of 3 items, total score will be calculated. To answer each question, five Likert-boxes were used (no pain, mild, moderate, severe, very severe). The average of the total scores of the patients in each arm will be provided.
PROMIS v1.0 Pain Intensity 3a Questionnaire Score | 2 weeks after surgery
  PROMIS is a computer adaptive test with branching logic. The Pain Intensity Questionnaire is comprised of 3 items, total score will be calculated. To answer each question, five Likert-boxes were used (no pain, mild, moderate, severe, very severe). The average of the total scores of the patients in each arm will be provided.
PROMIS v1.2 Physical Function Questionnaire Score | Baseline preoperatively
  PROMIS is a computer adaptive test with branching logic. The Physical Function Questionnaire is comprised of 170 items, total score will be calculated. To answer each question, five Likert-boxes were used (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). The average of the total scores of the patients in each arm will be provided.
PROMIS v1.2 Physical Function Questionnaire Score | 2 weeks after surgery
  PROMIS is a computer adaptive test with branching logic. The Physical Function Questionnaire is comprised of 170 items, total score will be calculated. To answer each question, five Likert-boxes were used (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). The average of the total scores of the patients in each arm will be provided.
PROMIS v2.0 Ability to Participate Socially Questionnaire Score | Baseline preoperatively
  PROMIS is a computer adaptive test with branching logic. The Ability to Participate Socially Questionnaire is comprised of 35 items, total score will be calculated. To answer each question, five Likert-boxes were used (never, rarely, sometimes, usually, always). The average of the total scores of the patients in each arm will be provided.
PROMIS v2.0 Ability to Participate Socially Questionnaire Score | 2 weeks after surgery
  PROMIS is a computer adaptive test with branching logic. The Ability to Participate Socially Questionnaire is comprised of 35 items, total score will be calculated. To answer each question, five Likert-boxes were used (never, rarely, sometimes, usually, always). The average of the total scores of the patients in each arm will be provided.
PROMIS v2.0 Satisfaction with Roles and Activities Questionnaire Score | Baseline preoperatively
  PROMIS is a computer adaptive test with branching logic. The Ability to Participate Socially Questionnaire is comprised of 44 items, total score will be calculated. To answer each question, five Likert-boxes were used (not at all, a little bit, somewhat, quite a bit, very much). The average of the total scores of the patients in each arm will be provided.
PROMIS v2.0 Satisfaction with Roles and Activities Questionnaire Score | 2 weeks after surgery
  PROMIS is a computer adaptive test with branching logic. The Ability to Participate Socially Questionnaire is comprised of 44 items, total score will be calculated. To answer each question, five Likert-boxes were used (not at all, a little bit, somewhat, quite a bit, very much). The average of the total scores of the patients in each arm will be provided.

OTHER OUTCOMES:
Time to Discharge | Up to 1 day (day of surgery)
  The average time for the experimental patients to be discharged (in minutes)
Percentage of patients reporting falls in the first 24 hours after surgery | 24 hours after surgery
  Falls will be self reported by patients

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Lynch, M.D., Principal Investigator — Columbia University Department of Orthopedics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] La Colla L, Ben-David B, Merman R. Quadratus Lumborum Block as an Alternative to Lumbar Plexus Block for Hip Surgery: A Report of 2 Cases. A A Case Rep. 2017 Jan 1;8(1):4-6. doi: 10.1213/XAA.0000000000000406. PMID 28036319
- [Background] La Colla L, Uskova A, Ben-David B. Single-shot Quadratus Lumborum Block for Postoperative Analgesia After Minimally Invasive Hip Arthroplasty: A New Alternative to Continuous Lumbar Plexus Block? Reg Anesth Pain Med. 2017 Jan/Feb;42(1):125-126. doi: 10.1097/AAP.0000000000000523. No abstract available. PMID 27997495
- [Background] Ben-David B, La Colla L. Extravasated Fluid in Hip Arthroscopy and Pain: Is Quadratus Lumborum Block the Answer? Anesth Analg. 2017 Jul;125(1):364. doi: 10.1213/ANE.0000000000002198. No abstract available. PMID 28609336